CLINICAL TRIAL: NCT04242862
Title: Study of the Prevalence, Risk Factors and Protective Factors of Burnout Among General Practitioners in France
Brief Title: Burn Out Among Medical Family Doctors
Acronym: BOUM
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Clermont-Ferrand (Other)
Collaborators: UFR Médecine & Pharmacie - Université Clermont Auvergne (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2016 BOUM
Record Dates: First submitted 2020-01-22; First posted 2020-01-27 (Actual); Last update posted 2020-01-27 (Actual); Status verified 2020-01

CONDITIONS: Burnout, Professional; Mental Health Wellness 1; Anxiety; Depressive Disorder; Occupational Stress
Keywords: General Practitioners; Private Practice; Models, Organizational; Behavior and Behavior Mechanisms; Test Anxiety Scale; Surveys and Questionnaires; Cross-Sectional Studies
MeSH Terms: conditions — Burnout, Professional; Anxiety Disorders; Depressive Disorder; Occupational Stress; Behavior

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The main objective of this study is to assess the burnout prevalence among French general practitioners in private practice.

As secondary outcomes, this study aim to measure the impact of sociodemographic variables, organizational practice models and workload. the investigators also intend to characterize the prevalence of depression, anxiety, fatigue and stress, drugs and alcohol consumption, use of psychotropic medication, and preferred strategies to cope with their symptoms.

DETAILED DESCRIPTION:
The BOUM protocol is designed to provide a better understanding of the current burnout prevalence among French general practitioners, as well as its risk and protective factors.

In order to fulfil those objectives, the methodologist estimated a 1536 individuals sample size, using an expected prevalence of severe burnout ranged between 10% and 20% (from the the EGPRN study - Soler, J.K., et al., Burnout in European family doctors: the EGPRN study. Family Practice, 2008. 25(4): p. 245-265), thus allowing the investigators to retrieve results with a 95% confidence level and a 2% error margin.

All analyses will be performed in a bilateral formulation for a 5% alpha error under the Stata® software (version 13, StataCorp, College Station, US). A difference will be considered statistically significant for p<0.05. The population will be described as frequency and percentage for the categorical variables, and as mean ± standard deviation or median [interquartile range] for the quantitative variables, according to their statistical distribution (normality studied by the Shapiro-Wilk test). Confidence intervals for population prevalence will be characterised with a binomial test. Comparisons between groups of burnout will be performed using Chi2 or Fisher's exact test for the categorical variables (followed by a Marascuillo post-hoc tests if needed), and by an ANOVA or Kruskal-Wallis test if normality and homoscedasticity not respected (Bartlett test) for the quantitative variables (followed by Tukey-Kramer or Dunn tests when necessary). Finally, considering the variables clinically relevant and those with a pertinent univariate analysis results, a multivariate analyse of ordinal polynomial regression type will be proposed; its results will be expressed as relative risk with 95% confidence intervals and presented as a Forest-plot.

ELIGIBILITY:
Inclusion Criteria:

* General practitioners working in France

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: General practitioners working in France
Enrollment: 1536 (Estimated)
Dates: Start 2016-11-01 (Actual); Primary Completion 2021-06-01 (Estimated); Study Completion 2022-06-01 (Estimated)

PRIMARY OUTCOMES:
Burnout in French General Practitioners | Day 1
  To evaluate the burnout prevalence in French General Practitioners, using the Maslach Burn-Out Inventory questionnaire

SECONDARY OUTCOMES:
Anxiety | Day 1
  Hospital Anxiety and Depression scale will be assessed and related to with demographic information and occupational characteristics
Depression | Day 1
  Hospital Anxiety and Depression scalewill be assessed and related to with demographic information and occupational characteristics
Stress | Day 1
  Visual analog scale will be assessed and related to with demographic information and occupational characteristics
Fatigue | Day 1
  Visual analog scale will be assessed and related to with demographic information and occupational characteristics
sleep disturbance | Day 1
  Validated questionnaire will be assessed and related to with demographic information and occupational characteristics
Psychiatric history and clinical approaches | Day 1
  Participants will be asked about any previous psychiatric diagnosis, suicidal attempt, use of any psychotropic medication and usual stress management approaches.
Addictive behaviors | Day 1
  Alcohol, tobacco and other psychotropic drugs consumption, through questionnaires assessment

CONTACTS AND LOCATIONS:
Overall Officials: Frederic Dutheil, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU Clermont Ferrand, Clermont-Ferrand, Auvergne, France